CLINICAL TRIAL: NCT06265766
Title: Brain STimulation for Arm Recovery After Stroke 2
Acronym: B-STARS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jord Vink (Other)
Responsible Party: Sponsor-Investigator, Jord Vink, dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL85511.041.24; 85511 (Other: ABR number)
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Transcranial magnetic stimulation; Continuous theta burst stimulation; Upper limb recovery; TMS; cTBS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sham cTBS treatment is delivered with a sham TMS-coil.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active cTBS (Experimental): Active cTBS delivered with an active TMS coil
  Interventions: Device: Active cTBS
- Sham cTBS (Sham Comparator): Sham cTBS delivered with a sham TMS coil
  Interventions: Device: Sham cTBS

INTERVENTIONS:
Device: Active cTBS — 10 sessions of active cTBS delivered to the contralesional primary motor cortex, started within 3 weeks after stroke.
  Arms: Active cTBS
Device: Sham cTBS — 10 sessions of sham cTBS delivered to the contralesional primary motor cortex, started within 3 weeks after stroke.
  Arms: Sham cTBS

SUMMARY:
Rationale: Every year, about 40,000 people in the Netherlands have a stroke. After the initial admission to the hospital, about 15% of stroke survivors is admitted to a rehabilitation center because of remaining disabilities. Three out of four of these patients have upper limb dysfunction, hampering activities of daily living. Upper limb function plays a critical role in the performance of most daily life activities. In our phase II trial B-STARS, continuous theta burst stimulation (cTBS) treatment led to an absolute additional recovery of upper limb function of 17%, as measured with the Action Research Arm Test (ARAT) score three months after stroke. This improvement exceeds the minimal clinically important difference of 10%. cTBS treatment also resulted in a significant improvement in measures of activities and participation (of similar magnitude) and a reduction in the mean length of stay at the rehabilitation center by 18 days.

Objective: To assess the effectiveness and cost effectiveness of cTBS treatment in promoting upper limb recovery after stroke in patients admitted to a rehabilitation center.

Study design: A phase III, multi-center, double-blind, randomized, sham-controlled, clinical trial.

Study population: 454 patients aged 18 years or older with a first-ever ischemic stroke or intracerebral hemorrhage and a unilateral arm paresis, defined by a Motricity Index between 9 and 99, in whom cTBS treatment can be started within 3 weeks after stroke onset.

Intervention: 10 daily sessions of cTBS delivered over the contralesional primary motor cortex during a period of 2 weeks, delivered immediately before regular care physical therapy of the affected upper limb.

Main study parameters/endpoints: The primary endpoint will be the score on the upper extremity section of the Fugl-Meyer assessment (FM-UE) at 90 days after stroke. Secondary endpoints will include the score on the FM-UE at one year and the scores on the Action Research Arm Test, Nine Hole Peg Test, Stroke Impact Scale, EuroQol 5 Dimensions and modified Rankin Scale at 90 days and one year after stroke

ELIGIBILITY:
Inclusion Criteria:

* Age, 18 years or older
* First-ever unilateral ischemic stroke or intracerebral hemorrhage in a cerebral hemisphere or the brainstem;
* Unilateral upper limb paresis with a motricity index between 9 and 99;
* Possibility to start cTBS treatment within 21 days after stroke onset;
* Signed informed consent.

Exclusion Criteria:

* Upper limb paresis prior to stroke onset;
* Absolute contra-indication to TMS
* Magnetic sensitive objects implanted in the head or neck area (e.g. cochlear implants, implanted neurostimulator, pacemaker or defibrillator, metal splinters, metal fragments or metal clips);
* History of epilepsy;
* Other contra-indications that may potentially be harmful as determined by the treating rehabilitation physician;
* Severe impairments that can impede study participation as determined by the treating rehabilitation physician (i.e. extreme fatigue, severe communication deficits);
* Life expectancy shorter than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper extremity section of the Fugl-Meyer Assessment | at 90 days post-stroke
  The score ranges from 0 to 66 points with a higher score indicating better outcome

SECONDARY OUTCOMES:
Upper extremity section of the Fugl-Meyer Assessment | at 12 months post-stroke
  The score ranges from 0 to 66 points with a higher score indicating better outcome
Action Research Arm Test | at 90 days and 12 months post-stroke
  The score ranges from 0 to 57 points with a higher score indicating better outcome
modified Rankin Scale | at 90 days and 12 months post-stroke
  The score ranges from 0 to 6 points with a lower score indicating better outcome
Hand section of Stroke Impact Scale | at 90 days and 12 months post-stroke
  The score ranges from 0 to 25 points with a higher score indicating better outcome
Participation section of Stroke Impact Scale | at 90 days and 12 months post-stroke
  The score ranges from 0 to 40 points with a higher score indicating better outcome
EuroQol-5D | at 90 days and 12 months post-stroke
  The score ranges from 0 to 5 points per item with a higher score indicating better outcome
Nine Hole Peg Test | at 90 days and 12 months post-stroke
  The outcome ranges from 0 to 50 seconds with a shorter outcome indicating better outcome
Ipsilesional corticospinal excitability | within 12 hours after the 10th cTBS session
  Ipsilesional corticospinal excitability is defined as the resting motor threshold of the ipsilesional hemisphere as determined with single pulse TMS. The outcome ranges from 0 to 100% of the machine output
iMTA medical consumption questionnaire | at 6 and 12 months post-stroke
  This questionnaire aims to identify costs associated with medical consumption
iMTA productivity cost questionnaire | At 6 and 12 months post-stroke
  This questionnaire aims to identify costs associated with productivity loss of paid work.

CONTACTS AND LOCATIONS:
Locations (16):
- Netherlands (16):
  - Tolbrug, 's-Hertogenbosch
  - Reade, Amsterdam
  - Revalidatie Friesland, Beetsterzwaag
  - Revant, Breda
  - MRC Aardenburg, Doorn
  - Libra Blixembosch, Eindhoven
  - University Medical Center Groningen, Groesbeek
  - Merem, Hilversum
  - Adelante, Hoensbroek
  - Basalt, Leiden
  - Sint Maartenskliniek, Nijmegen
  - Basalt, The Hague
  - Libra Leijpark, Tilburg
  - De Hoogstraat, Utrecht
  - Heliomare, Wijk aan Zee
  - Vogellanden, Zwolle

IPD SHARING:
Plan to Share IPD: No
Anonymized patient data can be made available on request